CLINICAL TRIAL: NCT02555267
Title: Multi-center, Prospective Cohort Study to Investigate the Impact of Comprehensive Geriatric Assessments on Survival and Toxicities in Elderly Diffuse Large B-cell Lymphoma Patients Treated With R-CHOP
Brief Title: Geriatric Assessments in Elderly Diffuse Large B-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: The Catholic University of Korea (Other); Kyungpook National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Korea University Anam Hospital (Other); Korea University Guro Hospital (Other); Kosin University Gospel Hospital (Other); Pusan National University Hospital (Other); Soonchunhyang University Hospital (Other); Ajou University School of Medicine (Other); Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Ho-Young Yhim, Assistant professor, Chonbuk National University Hospital
Other Study IDs: GERIAD
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma, Large B-cell, Diffuse
Keywords: geriatric assessment; diffuse large B-cell lymphoma; activity of daily living; instrumental activity of daily living; Charlson's comorbidity index
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly patients with DLBCL: Elderly patients (age>=65 years) with DLBCL treated with R-CHOP chemotherapy

SUMMARY:
This study investigate the impact of comprehensive geriatric assessments using activity of daily living (ADL), instrumental activity of daily living (IADL), and Charlson's comorbidity index (CCI) on survival and toxicities in Korean patients with diffuse large B-cell lymphoma (DLBCL) treated with R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed CD20+ DLBCL
* 65 years old or over
* Scheduled to receive R-CHOP chemotherapy
* Informed consent

Exclusion Criteria:

* Other histology than CD20+ DLBCL
* Primary central nervous system DLBCL
* Patients with a diagnosis of cancer (other than basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, well differentiated thyroid cancer [papillary or follicular thyroid cancer]) within 3 years before the study entry or with any treatment for cancer within 3 years before entry
* Consent withdrawal

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (≥ 65 years) with DLBCL treated with R-CHOP
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 2 years
  Event-free survival was defined as death, relapse from complete remission, progression during or after treatment, and discontinuation or changes of therapy during treatments

SECONDARY OUTCOMES:
Overall survival | 5 years
Progression-free survival | 5 years
Cumulative incidence of grade 3/4 adverse events and premature treatment discontinuation | 1 year

OTHER OUTCOMES:
Average received relative dose intensity | 6 months
  The dose intensity of each agent of R-CHOP chemotherapy was calculated by dividing the total received dose of the agent by the number of weeks of treatment. The relative dose intensity of each agents then was calculated by dividing the received dose intensity by the projected dose intensity for the agent. The sum of the relative dose intensities of the individual agents was divided by the number of agents in the R-CHOP to yield the average received relative dose intensity. In this study the average received relative dose intensity is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Young Yhim, MD, PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea